CLINICAL TRIAL: NCT01358578
Title: A Randomized, Double-blind, Double-dummy, Placebo Controlled, Multicenter Study of Subcutaneous Secukinumab to Demonstrate Efficacy After Twelve Weeks of Treatment, Compared to Placebo and Etanercept, and to Assess the Safety, Tolerability and Long-term Efficacy up to One Year in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Safety and Efficacy of Secukinumab Compared to Etanercept in Subjects With Moderate to Severe, Chronic Plaque-Type Psoriasis
Acronym: FIXTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2303; 2010-022228-66
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Results first posted 2015-09-23 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis,; inflammatory skin disease,; scaly patches; Psoriasis; inflammatory skin disease
MeSH Terms: conditions — Psoriasis; Dermatitis | interventions — secukinumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AIN457 150mg (Experimental): AIN457 150mg
  Interventions: Drug: Placebo; Drug: secukinumab (AIN457)
- AIN457 300mg (Experimental): AIN457 300mg
  Interventions: Drug: Placebo; Drug: secukinumab (AIN457)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Etanercept (Active Comparator): Etanercept
  Interventions: Drug: Placebo; Drug: etanercept
- AIN457 150mg from Placebo (Experimental): Patients randomized to AIN457 150mg in Maintenance phase when they were on Placebo in Induction Phase
  Interventions: Drug: Placebo; Drug: secukinumab (AIN457)
- AIN457 300mg from Placebo (Experimental): Patients randomized to AIN457 300mg in Maintenance phase when they were on Placebo in Induction Phase
  Interventions: Drug: Placebo; Drug: secukinumab (AIN457)

INTERVENTIONS:
Drug: Placebo — Placebo to Match secukinumab (AIN457) 150mg or 300mg or Placebo to match etanercept
Drug: secukinumab (AIN457) — secukinumab (AIN457) 150mg or 300mg subcutaneous
  Arms: AIN457 150mg; AIN457 150mg from Placebo; AIN457 300mg; AIN457 300mg from Placebo
Drug: etanercept — etanercept 50mg subcutaneous
  Arms: Etanercept

SUMMARY:
This study will assess the safety and efficacy of secukinumab compared to placebo and etanercept in patients that have moderate to severe, chronic, plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic, plaque-type psoriasis for at least 6 months
* Must have moderate to severe psoriasis based on PASI greater than 12, IGA greater than 3, and greater than 10% body surface area
* Must be inadequately controlled by prior treatments (topicals, phototherapy, and/or systemic therapies)

Exclusion Criteria:

* Forms of psoriasis other than chronic, plaque-type (such as pustular, erythrodermic and guttate psoriasis)
* Drug induced psoriasis
* Use of other psoriasis treatments during the study
* Prior use of etanercept
* Prior use of secukinumab or any other drug that target IL-17 (interleukin 17) or the IL-17 receptor
* Pregnant or lactating women; women who do not agree to use contraception during the study and for 16 weeks after stopping treatment
* Significant medical problems such as uncontrolled high blood pressure, congestive heart failure, etc.
* History of an ongoing, chronic or recurrent infection or evidence of tuberculosis
* Allergy to rubber or latex

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (128):
- United States (12):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Warren, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Johnston, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Norfolk, Virginia
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Carlton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Canada (8):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Richmond Hil, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Colombia (3):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Novartis Investigative Site, Alexandria, Egypt
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Turku
- France (7):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
- Germany (31):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wuppertal
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Kopavogur, Iceland
- India (9):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Dadar (east) Mumbai, Maharashtra
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Dehli, New Delhi
  - Novartis Investigative Site, Hyderabad
- Italy (7):
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Terracina, LT
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Philippines (2):
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Manila
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Singapore, Singapore
- South Korea (6):
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santa Coloma de Gramanet, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Uppsala
- United Kingdom (7):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Dudley
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nuneaton

REFERENCES:
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Houghton K, Patil D, Gomez B, Feldman SR. Correlation Between Change in Psoriasis Area and Severity Index and Dermatology Life Quality Index in Patients with Psoriasis: Pooled Analysis from Four Phase 3 Clinical Trials of Secukinumab. Dermatol Ther (Heidelb). 2021 Aug;11(4):1373-1384. doi: 10.1007/s13555-021-00564-2. Epub 2021 Jun 10. PMID 34110605
- [Derived] Dehlin M, Fasth AER, Reinhardt M, Jacobsson LTH. Impact of psoriasis disease activity and other risk factors on serum urate levels in patients with psoriasis and psoriatic arthritis-a post-hoc analysis of pooled data from three phase 3 trials with secukinumab. Rheumatol Adv Pract. 2021 Feb 18;5(1):rkab009. doi: 10.1093/rap/rkab009. eCollection 2021. PMID 33748660
- [Derived] Augustin M, Thaci D, Eyerich K, Pinter A, Radtke M, Lauffer F, Mrowietz U, Gerdes S, Pariser D, Lebwohl M, Sieder C, Melzer N, Reich K. Continued treatment with secukinumab is associated with high retention or regain of response. Br J Dermatol. 2020 Jan;182(1):67-75. doi: 10.1111/bjd.17991. Epub 2019 Jul 17. PMID 30972746
- [Derived] Menter A, Cather JC, Jarratt M, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab on Moderate-to-severe Plaque Psoriasis Affecting Different Body Regions: a Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):639-647. doi: 10.1007/s13555-016-0140-7. Epub 2016 Aug 30. PMID 27576559
- [Derived] Kircik L, Fowler J, Weiss J, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab for Moderate-to-Severe Head and Neck Psoriasis Over 52 Weeks: Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):627-638. doi: 10.1007/s13555-016-0139-0. Epub 2016 Aug 30. PMID 27573260
- [Derived] Gottlieb AB, Langley RG, Philipp S, Sigurgeirsson B, Blauvelt A, Martin R, Papavassilis C, Mpofu S. Secukinumab Improves Physical Function in Subjects With Plaque Psoriasis and Psoriatic Arthritis: Results from Two Randomized, Phase 3 Trials. J Drugs Dermatol. 2015 Aug;14(8):821-33. PMID 26267726
- [Derived] Langley RG, Elewski BE, Lebwohl M, Reich K, Griffiths CE, Papp K, Puig L, Nakagawa H, Spelman L, Sigurgeirsson B, Rivas E, Tsai TF, Wasel N, Tyring S, Salko T, Hampele I, Notter M, Karpov A, Helou S, Papavassilis C; ERASURE Study Group; FIXTURE Study Group. Secukinumab in plaque psoriasis--results of two phase 3 trials. N Engl J Med. 2014 Jul 24;371(4):326-38. doi: 10.1056/NEJMoa1314258. Epub 2014 Jul 9. PMID 25007392
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=56

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 150mg: s.c. secukinumab 150 mg injection plus a placebo secukinumab injection once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks, starting at Week 4, and until Week 48
- AIN457 300mg: s.c. secukinumab 300 mg injection plus a placebo secukinumab injection once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks, starting at Week 4, and until Week 48
- Placebo: s.c. placebo etanercept twice per week until Week 12 and s.c. placebo secukinumab (2 injections per dose) once per week for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks (at Weeks 4 and 8). Prior to receiving the Week 12 dose, all patients in the placebo group were assigned to the following treatment groups based on their PASI 75 response status at Week 12:
- Etanercept: Subcutaneous (s.c.) etanercept 50 mg twice per week until Week 12, followed by s.c. etanercept 50 mg every week from Week 12 through Week 51. To maintain the blind, patients also received 2 placebo secukinumab s.c.
  injections once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks, starting at Week 4, and until Week 48, except for Weeks 13, 14, and 15 where patients received an additional weekly dose (comprised of 2 s.c. injections per dose) of placebo secukinumab.
- AIN457 150mg From Placebo: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12 were re randomized to AIN457 150 in maintenance
- AIN457 300mg From Placebo: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12 were re randomized to AIN457 300 in maintenance
Period: Induction Period
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Etanercept | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 327 | 327 | 326 | 326 | 0 (These groups are populated after the induction period) | 0 (These groups are populated after the induction period)
Completed | 315 | 312 | 301 | 305 | 0 (These groups are populated after the induction period) | 0 (These groups are populated after the induction period)
Not Completed | 12 | 15 | 25 | 21 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 2 | 6 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 9 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 4 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 3 | 5 | 0 | 3 | 0 | 0
Not completed — technical problems | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 10 | 6 | 0 | 0
Period: Maintenance Period
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Etanercept | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 315 | 312 | 17 | 305 | 142 | 142
Completed | 276 | 290 | 15 | 263 | 125 | 131
Not Completed | 39 | 22 | 2 | 42 | 17 | 11
Not completed — Adverse Event | 2 | 7 | 0 | 6 | 4 | 3
Not completed — Lack of Efficacy | 10 | 2 | 0 | 11 | 3 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 5 | 1 | 1
Not completed — Non-compliance with study treatment | 3 | 1 | 0 | 2 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 7 | 4 | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 12 | 7 | 2 | 15 | 6 | 3
Period: Follow-up Period
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Etanercept | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 148 (Patients prior to follow up who did not enter the extension study but received the 150 mg dose) | 125 (Patients prior to follow up who did not enter the extension study but received the 300 mg dose) | 26 (contains patients who participated in follow up period from induction and maintenance) | 279 (contains patients who participated in follow up period from induction and maintenance) | 0 (all placebo patients from induction were 1: 1 into either AIN457A 150 mg or 300 mg doses) | 0 (all placebo patients from induction were 1: 1 into either AIN457A 150 mg or 300 mg doses)
Completed | 138 | 119 | 21 (contains patients who completed follow up period from induction and maintenance) | 260 (contains patients who completed follow up period from induction and maintenance) | 0 (all placebo patients from induction were 1: 1 into either AIN457A 150 mg or 300 mg doses) | 0 (all placebo patients from induction were 1: 1 into either AIN457A 150 mg or 300 mg doses)
Not Completed | 10 | 6 | 5 | 19 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 4 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 4 | 0 | 0
Not completed — non- compliance with study treatment | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 12 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Etanercept | Total
Number analyzed (Participants) | 327 | 327 | 326 | 326 | 1306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 304 | 305 | 311 | 308 | 1228
  >=65 years | 23 | 22 | 15 | 18 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (12.92) | 44.5 (13.19) | 44.1 (12.64) | 43.8 (12.95) | 44.4 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 103 | 89 | 94 | 377
  Male | 236 | 224 | 237 | 232 | 929
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 22 | 25 | 27 | 102
  Asian | 72 | 73 | 72 | 74 | 291
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 3
  Black or African American | 3 | 2 | 3 | 0 | 8
  White | 219 | 224 | 218 | 219 | 880
  More than one race | 5 | 5 | 5 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Secukinumab Compared to Placebo in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure: PASI 75 (Psoriasis Area and Severity Index) .
Description: A 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 75) is the current benchmark of primary endpoints for most clinical trials of psoriasis
Time Frame: 12 wks
Measure: Number; unit: participants achieving goal
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 327 | 323 | 324
participants achieving goal | 219 | 249 | 16

2. Primary Outcome: Efficacy of Secukinumab Compared to Placebo in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure:IGA (Investigator's Global Assessment) Mod 2011 With a 0 or 1 Response at Week 12
Description: The IGA mod 2011 scale has been developed based on a previous version of the scale used in secukinumab phase II studies in collaboration with health authorities, in particular the FDA. The explanations/descriptions of the points on the scale have been improved to ensure appropriate differentiation between the points. The IGA mod 2011 used in this study is static, i.e. it refers exclusively to the subject's disease state at the time of the assessments, and does not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit.IGA mod 2011 has a scale of 0-4 with the lower scores correlating to better performance. A score of 0= clear skin, 1= almost clear skin, 2=mild, 3=moderate,4=severe.
Time Frame: 12 wks
Measure: Number; unit: participants acheiving goal
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 327 | 323 | 324
participants acheiving goal | 167 | 202 | 9

3. Secondary Outcome: Efficacy of Secukinumab Compared to Etanercept and Placebo in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure: PASI 90 at Week 12
Description: A 90% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 90) is above current benchmark of primary endpoints for most clinical trials of psoriasis
Time Frame: 12 wks
Population: FAS
Measure: Number; unit: participant who acheived goal
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept | Placebo
Number analyzed (Participants) | 327 | 323 | 323 | 324
participant who acheived goal | 137 | 175 | 67 | 5

4. Secondary Outcome: Efficacy of Secukinumab Compared to Etanercept in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure: PASI 75 at Week 12
Description: as for outcome 1
Time Frame: 12 wks
Population: FAS
Measure: Number; unit: participant who acheived goal
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept
Number analyzed (Participants) | 327 | 323 | 323
participant who acheived goal | 219 | 249 | 142

5. Secondary Outcome: Efficacy of Secukinumab Compared to Etanercept in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Measure: :IGA (Investigator's Global Assessment) Mod 2011 With a 0 or 1 Response at Week 12
Description: as for outcome 2
Time Frame: 12 wks
Population: FAS
Measure: Number; unit: participant acheiving goal
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept
Number analyzed (Participants) | 327 | 323 | 323
participant acheiving goal | 167 | 202 | 88

6. Secondary Outcome: Maintenance of PASI 75 Response at Week 52 for Patients Who Were PASI 75 Responders at Week 12 (Non-responder Imputation)
Time Frame: 52 wks
Population: Full analysis set
Measure: Number; unit: participants who reached goal
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept
Number analyzed (Participants) | 219 | 249 | 142
participants who reached goal | 180 | 210 | 103

7. Secondary Outcome: Maintenance of IGA Mod 2011 0 or 1 Response After 52 Weeks of Treatment for Subjects Who Were IGA Mod 2011 0 or 1 Responders After 12 Weeks of Treatment
Time Frame: 52 wks
Population: Full analysis set
Measure: Number; unit: participants who reached goal
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept
Number analyzed (Participants) | 167 | 202 | 88
participants who reached goal | 113 | 161 | 50

8. Secondary Outcome: Change in Score From Baseline to Week 12 in Psoriasis Symptom Diary Items Itching, Pain and Scaling in AIN457 vs Placebo
Description: The Psoriasis Symptom Diary©, a 16-item patient reported outcome (PRO) measure developed and validated in accordance with the FDA PRO Guidance (FDA Guidance for Industry: Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims, 2009), demonstrated favorable psychometric properties and usefulness for treatment efficacy evaluation alongside other measures of disease severity in clinical trials for chronic plaque psoriasis.Weekly averages will be derived for each of the 16 questions of the Psoriasis Diary up to Week 12. A weekly average is the sum of the scored item over the course of the study week divided by the number of days on which the item was completed and will be set to missing if four or more daily assessments were missing of the corresponding question. The range for each question is 0 to 10 with the higher score depicting a more progressed disease state. A reduction in score from baseline shows efficacy
Time Frame: baseline to week 12
Population: Full analysis set
Measure: Mean (Standard Error); unit: units on scale
Groups:
- Placebo: AIN457A exact match Placebo
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 117 | 117 | 109
units on scale
  Itching | -4.92 (0.249) | -4.93 (0.247) | -0.54 (0.201)
  Pain | -4.10 (0.277) | -4.48 (0.278) | -0.33 (0.216)
  Scaling | -4.89 (0.241) | -4.93 (0.258) | -0.42 (0.217)

9. Secondary Outcome: Change From Baseline to Week 12 in Psoriasis Symptom Diary Items Itching, Pain and Scaling in AIN457 vs Etanercept
Description: as for outcome 8
Time Frame: baseline to week 12
Population: Full analysis set
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Etanercept: etanercept 50 mg twice per week until Week 12
Arm/Group | AIN457 150mg | AIN457 300mg | Etanercept
Number analyzed (Participants) | 117 | 117 | 116
Units on a scale
  Itching | -4.92 (0.277) | -4.93 (0.278) | -3.80 (0.257)
  Pain | -4.10 (0.268) | -4.48 (0.269) | -3.48 (0.251)
  Scaling | -4.89 (0.241) | -4.93 (0.258) | -3.74 (0.260)

10. Secondary Outcome: Number of Participants Developing Anti-secukinumab Antibodies
Description: Describes the number of participants tested positive for anti-secukinumab antibodies. It refers to the number of patients who had no positive values at baseline but developed them only after start of active study treatment (AIN457 or etanercept)
Time Frame: 60 weeks
Population: Full Analysis Set
Measure: Number; unit: # participants tested positive
Groups:
- PLACEBO-150 mg AIN457: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12 were re randomized to AIN457 150 in maintenance
- PLACEBO-300 mg AIN457: Patients were on Placebo in induction phase and if they were PASI 75 non responders at week 12 were re randomized to AIN457 300 in maintenance
- Placebo: s.c. placebo etanercept twice per week until Week 12 and s.c. placebo secukinumab (2 injections per dose) once per week for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks (at Weeks 4 and 8). Prior to receiving the Week 12 dose, all patients in the placebo group were assigned to treatment groups based on their PASI 75 response status at Week 12:
Arm/Group | AIN457 150mg | AIN457 300mg | PLACEBO-150 mg AIN457 | PLACEBO-300 mg AIN457 | Placebo | Etanercept
Number analyzed (Participants) | 327 | 327 | 142 | 142 | 17 | 326
# participants tested positive | 2 | 3 | 0 | 0 | 0 | 6

ADVERSE EVENTS:
Groups:
- INDUCTION-AIN457 150mg: INDUCTION-AIN457 150mg
- INDUCTION-AIN457 300mg: INDUCTION-AIN457 300mg
- INDUCTION-Placebo: INDUCTION-Placebo
- INDUCTION-Etanercept: INDUCTION-Etanercept
- ENTIRE-AIN457 150mg: ENTIRE-AIN457 150mg
- ENTIRE-AIN457 300mg: ENTIRE-AIN457 300mg
- ENTIRE-Any AIN457 150mg: ENTIRE-Any AIN457 150mg
- ENTIRE-Any AIN457 300mg: ENTIRE-Any AIN457 300mg
- ENTIRE-Placebo: ENTIRE-Placebo
- ENTIRE-Etanercept: ENTIRE-Etanercept
- FOLLOW UP-Any AIN457 150mg: FOLLOW UP-Any AIN457 150mg
- FOLLOW UP-Any AIN457 300mg: FOLLOW UP-Any AIN457 300mg
- FOLLOW UP-Placebo: FOLLOW UP-Placebo
- FOLLOW UP-Etanercept: FOLLOW UP-Etanercept
Arm/Group | INDUCTION-AIN457 150mg | INDUCTION-AIN457 300mg | INDUCTION-Placebo | INDUCTION-Etanercept | ENTIRE-AIN457 150mg | ENTIRE-AIN457 300mg | ENTIRE-Any AIN457 150mg | ENTIRE-Any AIN457 300mg | ENTIRE-Placebo | ENTIRE-Etanercept | FOLLOW UP-Any AIN457 150mg | FOLLOW UP-Any AIN457 300mg | FOLLOW UP-Placebo | FOLLOW UP-Etanercept
Serious Adverse Events (participants affected / at risk) | 7/327 | 4/326 | 6/327 | 3/323 | 18/327 | 21/326 | 24/469 | 27/467 | 7/327 | 20/323 | 2/148 | 2/125 | 0/27 | 2/278
Other Adverse Events (participants affected / at risk) | 157/327 | 145/326 | 121/327 | 130/323 | 225/327 | 230/326 | 297/469 | 316/467 | 122/327 | 213/323 | 25/148 | 11/125 | 7/27 | 59/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=327) | INDUCTION-AIN457 300mg (N=326) | INDUCTION-Placebo (N=327) | INDUCTION-Etanercept (N=323) | ENTIRE-AIN457 150mg (N=327) | ENTIRE-AIN457 300mg (N=326) | ENTIRE-Any AIN457 150mg (N=469) | ENTIRE-Any AIN457 300mg (N=467) | ENTIRE-Placebo (N=327) | ENTIRE-Etanercept (N=323) | FOLLOW UP-Any AIN457 150mg (N=148) | FOLLOW UP-Any AIN457 300mg (N=125) | FOLLOW UP-Placebo (N=27) | FOLLOW UP-Etanercept (N=278)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BASEDOW'S DISEASE (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PARATHYROID GLAND ENLARGEMENT (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THYROTOXIC CRISIS (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
POLYSEROSITIS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL HYPOTHYROIDISM (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TENDON INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FACIAL PARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VITH NERVE PARALYSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRUG ABUSE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CALCULUS URETHRAL (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LICHEN SCLEROSUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
ABSTAINS FROM ALCOHOL (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
BEHCET'S SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=327) | INDUCTION-AIN457 300mg (N=326) | INDUCTION-Placebo (N=327) | INDUCTION-Etanercept (N=323) | ENTIRE-AIN457 150mg (N=327) | ENTIRE-AIN457 300mg (N=326) | ENTIRE-Any AIN457 150mg (N=469) | ENTIRE-Any AIN457 300mg (N=467) | ENTIRE-Placebo (N=327) | ENTIRE-Etanercept (N=323) | FOLLOW UP-Any AIN457 150mg (N=148) | FOLLOW UP-Any AIN457 300mg (N=125) | FOLLOW UP-Placebo (N=27) | FOLLOW UP-Etanercept (N=278)
CONJUNCTIVITIS (Eye disorders) | 0 | 3 | 1 | 0 | 3 | 9 | 3 | 10 | 1 | 3 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 3 | 4 | 3 | 7 | 5 | 11 | 6 | 4 | 8 | 1 | 0 | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 2 | 4 | 1 | 10 | 10 | 12 | 14 | 4 | 3 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 12 | 17 | 6 | 11 | 30 | 34 | 36 | 38 | 7 | 22 | 2 | 1 | 0 | 3
NAUSEA (Gastrointestinal disorders) | 6 | 8 | 7 | 4 | 10 | 9 | 10 | 11 | 7 | 7 | 1 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 3 | 6 | 5 | 3 | 10 | 10 | 12 | 13 | 6 | 7 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 4 | 1 | 5 | 2 | 10 | 4 | 10 | 1 | 9 | 0 | 0 | 0 | 1
ADVERSE DRUG REACTION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 5 | 7 | 3 | 5 | 9 | 14 | 12 | 16 | 3 | 6 | 0 | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 2 | 1 | 3 | 7 | 5 | 7 | 8 | 1 | 9 | 1 | 1 | 0 | 1
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 5 | 1 | 4 | 1 | 9 | 3 | 10 | 4 | 4 | 5 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 2 | 5 | 3 | 7 | 10 | 12 | 14 | 19 | 3 | 15 | 1 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 4 | 4 | 2 | 4 | 12 | 15 | 14 | 17 | 2 | 9 | 0 | 0 | 0 | 2
EAR INFECTION (Infections and infestations) | 0 | 1 | 1 | 0 | 4 | 8 | 4 | 8 | 1 | 1 | 0 | 0 | 0 | 1
FOLLICULITIS (Infections and infestations) | 4 | 0 | 1 | 3 | 9 | 9 | 14 | 13 | 1 | 8 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 3 | 5 | 2 | 3 | 10 | 15 | 12 | 18 | 3 | 8 | 0 | 0 | 0 | 0
IMPETIGO (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 7 | 1 | 9 | 0 | 1 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 5 | 5 | 3 | 2 | 9 | 18 | 12 | 22 | 3 | 11 | 0 | 0 | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 44 | 35 | 26 | 37 | 82 | 91 | 107 | 122 | 26 | 87 | 6 | 1 | 3 | 14
ORAL CANDIDIASIS (Infections and infestations) | 1 | 2 | 0 | 0 | 4 | 10 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 1 | 5 | 0 | 0 | 1 | 8 | 4 | 10 | 0 | 9 | 0 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 5 | 4 | 0 | 0 | 7 | 9 | 10 | 13 | 0 | 6 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 4 | 7 | 4 | 3 | 7 | 10 | 8 | 14 | 4 | 6 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 5 | 0 | 1 | 0 | 9 | 8 | 11 | 9 | 1 | 5 | 0 | 0 | 0 | 1
TINEA PEDIS (Infections and infestations) | 3 | 3 | 0 | 0 | 6 | 8 | 7 | 10 | 0 | 4 | 0 | 0 | 0 | 0
TONSILLITIS (Infections and infestations) | 3 | 2 | 2 | 0 | 7 | 9 | 10 | 12 | 2 | 3 | 0 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 1 | 4 | 2 | 1 | 3 | 0 | 0 | 1 | 0
TRICHOMONIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 7 | 3 | 7 | 21 | 19 | 26 | 26 | 3 | 18 | 0 | 0 | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 2 | 2 | 3 | 6 | 6 | 8 | 8 | 13 | 3 | 9 | 1 | 0 | 0 | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 1 | 0 | 7 | 7 | 8 | 11 | 1 | 1 | 2 | 0 | 0 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 0 | 9 | 3 | 9 | 3 | 3 | 0 | 0 | 0 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 6 | 1 | 5 | 4 | 10 | 5 | 10 | 6 | 5 | 7 | 2 | 0 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0 | 8 | 3 | 8 | 5 | 2 | 4 | 1 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 6 | 1 | 3 | 2 | 8 | 3 | 8 | 3 | 3 | 3 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 | 5 | 10 | 12 | 25 | 18 | 32 | 23 | 10 | 22 | 3 | 0 | 0 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 8 | 6 | 10 | 17 | 22 | 20 | 30 | 6 | 27 | 0 | 0 | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 10 | 3 | 10 | 4 | 1 | 1 | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 3 | 5 | 7 | 9 | 10 | 4 | 9 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 8 | 3 | 8 | 4 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 1 | 5 | 12 | 8 | 13 | 4 | 4 | 2 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 16 | 30 | 23 | 23 | 34 | 47 | 46 | 59 | 24 | 40 | 3 | 2 | 0 | 2
PARAESTHESIA (Nervous system disorders) | 2 | 1 | 2 | 1 | 7 | 4 | 7 | 5 | 2 | 3 | 2 | 0 | 0 | 0
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 4 | 4 | 13 | 24 | 16 | 30 | 4 | 12 | 1 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 7 | 4 | 15 | 21 | 19 | 26 | 7 | 10 | 0 | 1 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1 | 2 | 3 | 9 | 3 | 10 | 1 | 2 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1 | 8 | 9 | 10 | 11 | 0 | 2 | 0 | 0 | 0 | 3
ERYTHRODERMIC PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 4 | 1 | 4 | 1 | 0 | 2 | 3 | 5 | 0 | 12
PRURITUS (Skin and subcutaneous tissue disorders) | 12 | 8 | 11 | 9 | 18 | 14 | 21 | 17 | 11 | 16 | 2 | 1 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 5 | 1 | 7 | 2 | 9 | 5 | 11 | 7 | 7 | 6 | 2 | 0 | 0 | 5
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 7 | 5 | 8 | 5 | 0 | 2 | 0 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 2 | 7 | 3 | 9 | 4 | 0 | 3 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 10 | 5 | 4 | 5 | 18 | 16 | 22 | 20 | 4 | 14 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.